CLINICAL TRIAL: NCT04052919
Title: Cardiac Dysfunction in Adolescents With Type 1 Diabetes: Contribution of Daily-life Glucoregulation and Impact on Cardiorespiratory Exercise Capacity
Acronym: GIIADMT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Dominique Hansen, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GIIADMT1
Record Dates: First submitted 2017-12-19; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac dysfunction in adolescents with type 1 diabetes (Experimental): to identify specific parameters related to glucoregulation which correlate with cardiac function and structure in adolescent with T1DM.
  In T1DM, exercise training to have beneficial effects on HbA1c levels, cardiovascular risk profile.
  To evaluate the association between cardiac function/structure and cardiopulmonary exercise capacity in adolescent T1DM patients (in the perspective of their physical activity behavior). This study thus may provide greater insights in the etiology and consequences of a disturbed cardiac function/structure in adolescents with T1DM.
  Interventions: Other: Cardiac dysfunction in adolescents with type 1 diabetes

INTERVENTIONS:
Other: Cardiac dysfunction in adolescents with type 1 diabetes — to identify specific parameters related to glucoregulation which correlate with cardiac function and structure in adolescent with T1DM.
  In T1DM, exercise training to have beneficial effects on HbA1c levels, cardiovascular risk profile.
  To evaluate the association between cardiac function/structure and cardiopulmonary exercise capacity in adolescent T1DM patients (in the perspective of their physical activity behavior). This study thus may provide greater insights in the etiology and consequences of a disturbed cardiac function/structure in adolescents with T1DM.

SUMMARY:
During the course of type 1 diabetes mellitus (T1DM), several complications can occur. One of these is the development of diastolic and systolic dysfunction (even in the absence of ischemic, valvular or hypertensive heart disease). Such cardiac dysfunction and adverse remodeling is more common in adolescents with T1DM with a worse glycemic control (as evidenced by higher blood glycated hemoglobin HbA1c) concentrations. Even though an association has been observed between higher blood HbA1c concentrations and a worse cardiac function/structure in adolescents with T1DM, less is known about the specific characteristics of the glucoregulation (e.g. number and duration of hyperglycemic or hypoglycemic episodes, age of onset of T1DM,..) in relation to cardiac function/structure in this population. Therefore, the first aim of this study is to identify specific parameters related to glucoregulation which correlate with cardiac function and structure in adolescent with T1DM.

In T1DM, exercise training is generally recommended and included in the guidelines for the care of T1DM (due to beneficial effects on HbA1c levels, cardiovascular risk profile,..). However, as exercise training may increase the risk of hypoglycemic events, many patients may fear exercise, leading to inactivity or sedentarism. Logically, physical activity volumes are diverse in cohorts of this patient population, in which the long-term physically active T1DM patient will display an optimal or preserved cardiopulmonary exercise capacity, while a suboptimal cardiopulmonary exercise capacity will be noticed in mostly sedentary T1DM patients. The second aim of this study is to evaluate the association between cardiac function/structure and cardiopulmonary exercise capacity in adolescent T1DM patients (in the perspective of their physical activity behavior). This study thus may provide greater insights in the etiology and consequences of a disturbed cardiac function/structure in adolescents with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus

Exclusion Criteria:

* chronic diseases (except type 1 diabetes mellitus)
* disorders hindering exercise

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
transthoracic echocardiography | day 1
  cardiac function/structure via transthoracic echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)

SECONDARY OUTCOMES:
glycemic control | daily (day 1- day 14)
  continuous monitoring/evaluation of glucose concentrations via glucose
body composition | day 1
  Evaluation of body composition via bio-electrical impedance analyses. Via this analysis, the amount of fat-free body mass and fat body mass is calculated.
HbA1C level | day 1
  Evaluation of glycemic control
BMI (Body Mass Index) | day 1
  Assessment of body composition using body mass index
Height | day 1
  Anthropometric assessment
weight | day 1
  Anthropometric assessment
Physical activity questionaire | daily (day 1 - day 14)
  Assessment of physical activity using a validated questionnaire (PAQ-A)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided